CLINICAL TRIAL: NCT01470248
Title: A Single Arm, Two-Stage Phase II Study of Arsenic Trioxide in Previously Treated Small Cell Lung Cancer
Brief Title: Study of Arsenic Trioxide in Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Cephalon (Industry); Teva Pharmaceuticals USA (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Taofeek K. Owonikoko, Associate Professor, Hematology/Medical Oncology, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00050301; WCI1988-11 (Other: Other); K23CA164015 (NIH)
Record Dates: First submitted 2011-10-25; First posted 2011-11-11 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer; Cancer of Lung; Pulmonary Cancer; Pulmonary Neoplasms; Carcinoma, Small Cell
Keywords: Lung Cancer; Carcinoma, small cell; Trisenox; Arsenic trioxide; phase II trial
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Small Cell | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arsenic Trioxide Treatment (Experimental): This is a single arm study. All patients will be treated with the investigational agent, Arsenic Trioxide, according to the dose and schedule indicated in the protocol.
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide — Drug will be given as a loading dose of 0.32mg/kg/day for 4 days in Week 1, followed by 0.25mg/kg/day twice per week for 5 weeks, followed by 2 weeks of rest, at which time response assessment will be performed. Patients will be restaged prior to the beginning of a new cycle, every 2 months on average. Maximum of 6 cycles of therapy will be administered in the absence of tumor progression or excessive side effects
  Other Names: Trisenox; ATO

SUMMARY:
The purpose of this study is to study the effect of an anticancer drug, Arsenic Trioxide, in patients with small cell lung cancer who have failed at least one standard chemotherapy regimen as well as patients who are unable to tolerate the standard treatment for their cancer. The investigators seek to establish the safety of and efficacy of Arsenic Trioxide in this patient group. The study will include up to 36 participants with small cell lung cancer.

The investigators want to find out what effects, good or bad, that the study drug has on your cancer. This study will also look at specific biomarkers in your blood and in the tumor tissue which may help the investigators to determine if the levels of these biomarkers are related to tumor response to treatment.

Arsenic Trioxide, also known by the brand name, Trisenox, is a chemotherapy drug approved by the Food and Drug Administration (FDA) for the treatment of a specific type of blood cancer called Acute Promyelocytic Leukemia. It works in part by making cancer cells become more mature thereby stopping them from growing in number and more likely to die off.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed small cell lung cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as > 10 mm with spiral CT scan.
* Patient must have failed or found to be intolerant of standard frontline platinum-based regimens. There is no limit on the number of prior regimens provided the patient meets all the other eligibility criteria.
* Adult patients 18 years or older. Because no dosing or adverse event data are currently available on the use of arsenic trioxide in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count > 1,500/mL
  * platelets > 100,000/mL
  * total bilirubin ≤ 1.5 X institutional upper limits of normal
  * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 X institutional upper limit of normal
  * creatinine ≤ 1.5 X institutional upper limits of normal OR
  * creatinine clearance > 40 mL/min/1.73 m² for patients with
  * creatinine levels above institutional normal.
* Negative serum pregnancy test within 48 hours before starting study treatment in women with childbearing potential
* Ability to understand and the willingness to sign a written informed consent document.
* No history of QTc prolongation syndrome or any other cardiac conduction abnormality evidenced by normal baseline EKG (QTc ≤ 450 in males and ≤ 470 in females)
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Need for treatment with chemotherapy (within 4 weeks; 6 weeks for nitrosoureas or mitomycin C); radiotherapy or biologic agents (within 2 weeks) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with uncontrolled symptomatic brain metastases. Patients with no known brain metastasis are not required to undergo screening prior to enrolment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to arsenic trioxide.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Trisenox is a category D agent with the potential to cause fetal harm. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Trisenox, breastfeeding should be discontinued if the mother is treated with Trisenox.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Trisenox. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who require ongoing treatment with any hematopoietic colony-stimulating growth factors (e.g., granulocyte-colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF]) ≤ 2 weeks prior to starting study drug.
* Patients who are currently receiving treatment with medication that has the potential to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* History of another malignancy within 3 years, except curatively treated basal cell carcinoma of the skin, ductal carcinoma in situ (DCIS), early stage prostate cancer without detectable prostate-specific antigen (PSA) or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Result] Owonikoko TK, Zhang G, Kim HS, Stinson RM, Bechara R, Zhang C, Chen Z, Saba NF, Pakkala S, Pillai R, Deng X, Sun SY, Rossi MR, Sica GL, Ramalingam SS, Khuri FR. Patient-derived xenografts faithfully replicated clinical outcome in a phase II co-clinical trial of arsenic trioxide in relapsed small cell lung cancer. J Transl Med. 2016 May 3;14(1):111. doi: 10.1186/s12967-016-0861-5. PMID 27142472
- See also: Winship Clinical Trials — https://winshipcancer.emory.edu/patient-care/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled through the thoracic medical oncology clinic of the Winship Cancer Institute of Emory University, between August 2011 and April 2014.
Period: Overall Study
Arm/Group | Arsenic Trioxide Treatment
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arsenic Trioxide Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.40 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Response rate (complete response [CR]+ partial response [PR]) was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  * Complete response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  * Partial response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Progressive disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 8 weeks
Population: Two patients were not analyzed because only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated were considered evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Arsenic Trioxide Treatment
Number analyzed (Participants) | 17
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 2
  Progressive disease | 15

2. Primary Outcome: Clinical Benefit Rate (CBR)
Description: Sum of complete response (CR), partial response (PR) and stable disease (SD) in patients eligible for efficacy analysis.
Time Frame: After completing at least 1 cycle (8 weeks) of treatment
Population: An alternative endpoint of clinical benefit rate was pre-specified in the event that the study failed to meet its overall response rate (ORR) endpoint either at the end of stage I accrual or at final analysis. However, this study met its endpoint. Please see primary outcome measure 1.
Arm/Group | Arsenic Trioxide Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Description: Defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Every 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Arsenic Trioxide Treatment
Number analyzed (Participants) | 17
weeks | 6.26 (3.9)

4. Secondary Outcome: Overall Survival
Description: Duration of time from enrollment on study until death
Time Frame: From enrolment till death on average up to 2 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Arsenic Trioxide Treatment
Number analyzed (Participants) | 17
months | 4.5 [2 to 7]

ADVERSE EVENTS:
Time Frame: Patients were followed until study closure or until death, whichever occurred first.
Arm/Group | Arsenic Trioxide Treatment
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arsenic Trioxide Treatment (N=19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arsenic Trioxide Treatment (N=19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Elevated creatinine (Renal and urinary disorders) | 1
Facial edema around eyes (Skin and subcutaneous tissue disorders) | 1
Generalized weakness (General disorders) | 1
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 3
Hypocalcemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 1
Increased alkaline phosphatase (Blood and lymphatic system disorders) | 1
Increased lipase (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes